CLINICAL TRIAL: NCT05318989
Title: Epigenetic Profile of Vaginal Epithelial Cells in Postmenopausal Women and as a Result of Local Hormone Therapy, Assessed on the Basis of the Analysis of DNA Methylation Level and Expression of TET 1-3 Genes in Terms of the Aging Process
Brief Title: Genetic Aspects of Vaginal Aging
Status: Completed | Type: Observational
Sponsor: Żelazna Medical Centre, LLC (Other)
Collaborators: Laboratory of Genetics and Human Genomics, University of Gdańsk (Unknown)
Responsible Party: Principal Investigator, Jacek Szymański, Jacek Szymański MD, PhD, Żelazna Medical Centre, LLC
Other Study IDs: 1
Record Dates: First submitted 2022-02-24; First posted 2022-04-08 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Genitourinary Agents
Keywords: vulvovaginal atrophy; genitourinary syndrome of menopause; aging; 5-hydroxymethylcytosine; 5-hmC; 5-methylcytosine; ten-eleven translocation; TET enzymes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — vaginal swabs, buccal swabs, vaginal wall samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Premenopausal women (PREM): Control group
- Postmenopausal women (POSMA): Test group A : postmenopausal women not treated with topical estrogens
- Postmenopausal women (POSMB): Test group B: postmenopausal women treated with topical estrogens

SUMMARY:
Life expectancy depends on a number of different factors, of which only about 20-30% are genetically determined. The overwhelming majority are non-genetic determinants. One of the proposed mechanisms explaining this aging phenomenon is related to epigenome variability. Epigenetic regulation is mainly based on cytosine methylation / demethylation in DNA and modification of histone proteins. DNA methylation, unlike modification of histone proteins, is a permanent change, the effects of which can be very distant, and the methylation patterns are fixed during subsequent cell divisions. This type of epigenetic modification plays an important role in a variety of cellular processes, such as differentiation, transformation and aging. The most commonly methylated are cytosines within two nucleotide sequences in DNA called CpG islands. Numerous studies confirm the age-related reduction in methylcitosine (5-mC) levels in both the nuclear and mitochondrial genome of cells in various tissues. The enzymes that catalyze this process belong to the family of methyltransferases (DNMTs). Cytosine methylation appears to be one of the key processes in tissue aging. Depending on the type of tissue and DNA region, there is an increase or decrease in cytosine methylation with age. The main process of both passive and active demethylation is the hydroxymethylation of methylcytosine leading to the formation of hydroxymethylcytosine (5-hmC). This process is of great importance in the regulation of gene expression. Three hydroxylases, TET 1-3 enzymes (ten-eleven translocation), take part in the 5mC hydroxylation process in mammalian cells. The resulting 5-hmC is an important intermediate in the process of DNA demethylation. The significant decrease in the level of CpG island methylation in the genome also seems to be of key importance. So far, the role of 5mC, and thus the activity of TET enzymes in the aging process, has not been clearly defined. Previous studies have shown that it can play an important role in the development and aging of the body. In a woman's life, the consequences of the aging process are most severely manifested during the menopause. The deficiency of sex hormones determines a number of processes also occurring in the lower urinary tract. Estrogens are an essential regulator of the physiological function of the vagina. 40-60% of postmenopausal women complain of atrophic changes in the vaginal epithelium (VVA - vulvovaginal atrophy). Vaginal topical estrogens are currently the "gold standard" in VVA therapy. The molecular mechanism of action of estrogens is based on their activation of the estrogen receptors ER-alpha and ER-beta located in the nuclear envelope of cells in target organs. After the ligand binds to the appropriate receptor, a cascade of signals activating the appropriate chromatin-binding transcription factors is triggered. As a result of this process, the expression of genes involved in the processes of proliferation, differentiation as well as apoptosis changes. Therefore, local administration of estrogens is the most effective in improving the physiological condition of the vaginal mucosa epithelium. The question arises, how do hormonal deficiencies appearing in the menopausal period affect epigenetic changes in the genome and, consequently, the modification of gene expression related to the aging processes of the organism? Does the use of hormone therapy affect the regulation of gene expression through changes in the level of genome methylation? Can the determination of the level of total methylation in vaginal mucosa cells serve as a marker of the advancement of the aging process? Additionally, will the assessment of the degree of demethylation of the genome of vaginal mucosa cells by analyzing the level of expression of genes encoding TET 1-3 enzymes and the total level of 5mC allow characterizing epigenetic changes occurring in menopausal women? Is it possible to identify specific genes whose methylation-dependent expression regulates aging? Obtaining answers to such questions may contribute to understanding the role of the epigenome in the aging process of cells, and opening up new possibilities for the implementation of more effective therapies. It is also crucial that the vaginal epithelium is generally not exposed to known environmental factors influencing the course of aging (e.g. UV radiation), and thus the observed epigenetic changes in vaginal epithelial cells should reflect the impact of hormonal disorders on the molecular mechanism of aging.

ELIGIBILITY:
Inclusion Criteria:

* informed consent of the patient
* patient's age> 18 years
* POP-Q < = II
* non-smoker
* without prior vaginal surgery

Exclusion Criteria:

* refusal to participate in the study
* POP-Q > II
* smoking
* internal diseases (diabetes, disorders of the thyroid gland, obesity, cancer, malnutrition, exhaustion)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population description: Women treated in Urogynecological Unit of St. Sophia Hospital in Warsaw (outpatients and hospitalized) who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
5-hmC content | 30 days
  - 5-hmC content and 5-mC increase in tissues with urogenital atrophy
TET expressiion | 30 days
  - TET expression in tissues with urogenital atrophy
Changes in the 5-hmC | 30 days
  - changes in the 5-hmC content and the 5-mC content in vaginal cells after hormone therapy (topical application of estrogens)
TET expression change | 30 days
  - TET expression change after hormone therapy

SECONDARY OUTCOMES:
Promoter methylation of specific genes involved in the aging process | 30 days
  - Methylome analysis to identify promoter methylation of specific genes involved in the aging process

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum Medyczne "ŻELAZNA", Warsaw, Poland

REFERENCES:
- [Background] Palma F, Volpe A, Villa P, Cagnacci A; Writing group of AGATA study. Vaginal atrophy of women in postmenopause. Results from a multicentric observational study: The AGATA study. Maturitas. 2016 Jan;83:40-4. doi: 10.1016/j.maturitas.2015.09.001. Epub 2015 Sep 14. PMID 26421474
- [Background] Borkowska J, Domaszewska-Szostek A, Kolodziej P, Wicik Z, Polosak J, Buyanovskaya O, Charzewski L, Stanczyk M, Noszczyk B, Puzianowska-Kuznicka M. Alterations in 5hmC level and genomic distribution in aging-related epigenetic drift in human adipose stem cells. Epigenomics. 2020 Mar;12(5):423-437. doi: 10.2217/epi-2019-0131. Epub 2020 Feb 7. PMID 32031421
- [Background] Truong TP, Sakata-Yanagimoto M, Yamada M, Nagae G, Enami T, Nakamoto-Matsubara R, Aburatani H, Chiba S. Age-Dependent Decrease of DNA Hydroxymethylation in Human T Cells. J Clin Exp Hematop. 2015;55(1):1-6. doi: 10.3960/jslrt.55.1. PMID 26105999
- [Background] Gorodeski GI. Aging and estrogen effects on transcervical-transvaginal epithelial permeability. J Clin Endocrinol Metab. 2005 Jan;90(1):345-51. doi: 10.1210/jc.2004-1223. Epub 2004 Oct 13. PMID 15483084
- [Background] Li D, Guo B, Wu H, Tan L, Lu Q. TET Family of Dioxygenases: Crucial Roles and Underlying Mechanisms. Cytogenet Genome Res. 2015;146(3):171-80. doi: 10.1159/000438853. Epub 2015 Aug 21. PMID 26302812